CLINICAL TRIAL: NCT00460759
Title: Pharmacokinetic Issues in the Use of Moxifloxacin Plus Rifapentine
Brief Title: Pharmacokinetic Issues of Moxifloxacin Plus Rifapentine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00007322
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Mycobacterium Tuberculosis
Keywords: Mycobacterium tuberculosis, rifapentine, moxifloxacin
MeSH Terms: interventions — Moxifloxacin; rifapentine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moxifloxacin and Rifapentine (Experimental)
  Interventions: Drug: Moxifloxacin; Drug: Rifapentine

INTERVENTIONS:
Drug: Moxifloxacin
Drug: Rifapentine

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (how a drug is absorbed, distributed, and eliminated by the body) of moxifloxacin alone versus moxifloxacin given with rifapentine. Researchers believe that understanding how these tuberculosis drugs interact when given together may help to determine the best drug treatment plan for use in future studies. Volunteers will take moxifloxacin daily by mouth for the first part of the study and then moxifloxacin in combination with rifapentine during the second part of the study. Sixteen healthy men and women will be recruited from Johns Hopkins University School of Medicine to volunteer for this study. They will be required to stay in the inpatient unit twice, each time for 84 hours. Study procedures will include having a tube placed in a vein to draw several blood samples over time. Volunteers will participate in the study for a maximum of 48 days, including screening and follow-up visits.

DETAILED DESCRIPTION:
New drugs are urgently needed to shorten the duration of tuberculosis (TB) treatment and to facilitate the delivery of directly observed therapy. Preliminary data indicates that a TB treatment regimen that includes moxifloxacin plus rifapentine may have excellent antituberculosis activity that could allow for shortening of total TB treatment duration. However, little is known about possible pharmacokinetic interactions between the two drugs in humans. More specifically, moxifloxacin is metabolized via glucuronide and sulfate conjugation to inactive metabolites. Given that rifapentine induces the activity of phase II enzymes including glucuronosyltransferase and sulphotransferase, it is possible that rifapentine may alter the pharmacokinetics of moxifloxacin. This study will be a prospective, phase I, single center pharmacokinetic study in healthy subjects. The trial will compare the pharmacokinetics of moxifloxacin alone versus moxifloxacin administered with thrice-weekly rifapentine, each administered orally. There will be two parts to the trial: Part I (Days 1-4) during which moxifloxacin is administered alone; and Part II (Days 5-19) during which moxifloxacin is co-administered with thrice-weekly rifapentine. A 24-hour pharmacokinetic profile of moxifloxacin will be obtained following dose administration of moxifloxacin on Day 4 to obtain baseline steady state data at a dose of 400 mg daily. On Day 5, rifapentine will be added to the regimen at a dose of 900 mg thrice weekly, and a 48-hour pharmacokinetic profile for rifapentine and its metabolite, 25-desacetyl-rifapentine will be obtained after the first dose. On Day 19, 72-hour pharmacokinetic profiles for moxifloxacin, rifapentine, and 25-desacetyl-rifapentine will be performed. Safety and tolerability assessments will be performed at designated intervals throughout the study. Beginning on Day 1, subjects will receive moxifloxacin 400 mg daily for 19 days (Days 1-19). Beginning on Day 5, subjects will also receive rifapentine 900 mg thrice weekly (to be administered on Days 5, 7, 9, 12, 14, 16 and 19). Study participants will be 16 healthy adults, ages 18-65, recruited through Johns Hopkins University School of Medicine. The primary study objectives are to: compare, in healthy volunteers, the pharmacokinetics of moxifloxacin alone versus moxifloxacin co-administered with thrice-weekly rifapentine and describe the safety and tolerability of moxifloxacin co-administered with rifapentine. The secondary study objective is to evaluate for rifapentine autoinduction of metabolism in healthy volunteers receiving thrice-weekly rifapentine. The primary safety outcome will be the proportion of subjects with any Grade 3 or 4 toxicity associated with study medications or any serious adverse event. The secondary safety outcomes will be the proportion of subjects with any Grade 1 or 2 toxicity associated with study medications, and the proportion of subjects discontinuing study medications for any reason.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* Age greater than or equal to 18 years, and less than or equal to 65 years.
* Within 14 or fewer days prior to enrollment, a complete blood count, comprehensive serum chemistry profile, and HIV antibody test will be performed, with the following laboratory values:
* Serum amino aspartate transferase (AST) at or within the normal limits for the laboratory
* Total bilirubin level at, below, or within the normal limits for the laboratory
* Creatinine level at, below, or within the normal limits for the laboratory
* Uric acid at, below, or within the normal limits for the laboratory
* Hemoglobin greater than 12.0 for men, greater than 11.0 for women
* Platelet count greater than or equal to 125,000/cu mm
* Absolute neutrophil count greater than or equal to 1250/cu mm
* Potassium level of at least 3.5 mEq/L
* Serum albumin at or within normal limits for the laboratory
* HIV antibody test negative
* For women of childbearing potential, a negative serum beta-Human Chorionic Gonadatropin (bHCG) pregnancy test, performed at screening and on Day 0.
* During the study and for 14 days after the last dose of study medication, women of childbearing potential must agree to practice a double-barrier method of birth control (e.g., condom plus spermicidal foam, condom plus diaphragm, etc) or to abstain from heterosexual vaginal intercourse since hormonal contraceptives will be prohibited during the study. Female subjects must plan on not getting pregnant during the study and for 14 days after the last dose of study medication.
* Access to a telephone for the duration of the study.
* Within 14 days or fewer prior to enrollment, an electrocardiogram with corrected QT interval (QTc) less than or equal to 0.44 seconds.

Exclusion Criteria:

* Breastfeeding
* Known intolerance to either of the study drugs or to fluoroquinolone antibiotics
* Use of rifamycin or fluoroquinolone antibiotics in the 30 days prior to enrollment
* Inability to take oral medications
* History of any renal, hepatic, cardiac (except benign heart murmur), or endocrine disorder; or malignancy; or immunocompromised
* History of any acute or chronic illness that requires current medical therapy
* Prior gastrointestinal surgery involving stomach, biliary system, pancreas, or small intestine
* Any medical condition that, in the opinion of the investigator, would interfere with the subject's ability to participate in the protocol
* Any illicit drug use within the preceding 2 months. Subjects must agree to abstain from alcohol, tobacco, and illicit drug use during the study
* Current use of any prescription medication(s)
* Planned use, during the study from Day 0 through the last PK blood draw, of any of the following: prescription medication(s), herbal supplement(s), vitamin(s), mineral supplement(s), or over-the-counter medication(s) with the exception of acetaminophen
* History of prolonged QT syndrome
* Participation in any other investigational drug study within 21 days prior to study entry and during the study
* Inability to participate in pharmacokinetic visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2008-08-24 (Actual); Study Completion 2008-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States